CLINICAL TRIAL: NCT05845398
Title: A Phase 1b, Double-blind, Placebo-controlled, Repeat-dose, Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Study of DCR-AUD in Healthy Volunteers
Brief Title: Phase 1b Study of DCR-AUD in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dicerna Pharmaceuticals, Inc., a Novo Nordisk company (Industry)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DCR-AUD-102
Record Dates: First submitted 2023-04-26; First posted 2023-05-06 (Actual); Results first posted 2025-01-03 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 3 to 1 to DCR-AUD or placebo.
Who Masked: Participant, Investigator
Masking Description: Participants and site study staff will be blinded to the randomization. Some members of the Sponsor team will be unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DCR-AUD (Experimental): Multiple doses of DCR-AUD. Subcutaneous administration of of DCR-AUD.
  Interventions: Drug: DCR-AUD
- DCR-AUD Placebo (Placebo Comparator): Multiple doses of placebo comparator. Subcutaneous administration of Placebo for DCR-AUD, volume to match active single dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DCR-AUD — DCR-A1203, the drug substance of DCR-AUD, is a synthetic double-stranded (hybridized duplex) RNA oligonucleotide conjugated to GalNAc ligands that enable specific hepatic access and update after subcutaneous administration. DCR-AUD is a sterile solution of DCR-A1203 at a concentration of 160 mg/mL in water for injection (WFI).
  Other Names: DCR-A1203
  Arms: DCR-AUD
Drug: Placebo — 0.9% saline for injection.
  Arms: DCR-AUD Placebo

SUMMARY:
The goal of this clinical trial is to test the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of of repeat doses of DCR-AUD in adult healthy volunteers who are social drinkers.

The main questions it aims to answer are:

* Are repeat doses of DCR-AUD safe and well-tolerated in healthy adults who are social drinkers?
* How does the drug behave inside the human body and how it is removed from the human body?
* What are the symptoms the drug may cause with alcohol consumption?

Participants will:

* Receive multiple doses of DCR-AUD.
* Have assessment visits through Week 24.
* Participate in up to 10 Ethanol Interaction Assessments (EIAs) to see how the body is affected by DCR-AUD.

Researchers will compare the groups of participates who receive study drug with the group of participants who receive placebo to see if the study drug is safe and tolerable and whether the study drug has any real effect.

ELIGIBILITY:
Inclusion Criteria:

1. 21 to 65 years, inclusive, at the time of signing informed consent.
2. Overtly healthy volunteers, as determined by medical evaluation including medical history, physical examination, and laboratory testing.
3. No diagnosis of AUD within the preceding 12 months per Diagnostic and Statistical Manual of Mental Disorders (DSM-5).
4. Social drinkers who consume, on average, 5 to 20 drinks per week for men or 5 to 14 drinks per week for women over the 4 weeks prior to Screening, and not more than 8 drinks in a single day.
5. No evidence of overt or sub-clinical hepatic pathology, as manifest by serologic tests demonstrating hepatic inflammation or compromised hepatic synthetic function (i.e., AST, ALT, GGT, total bilirubin < 1.5 times the ULN at Screening and Day -1).
6. eGFR ≥ 60 mL/min/1.73 m2 at Screening.
7. No history of significant adverse reaction(s) to alcohol. Participant should be expected to tolerate the amount of alcohol administered during EIAs.
8. Willing to participate in up to 10 EIAs.
9. Has a negative test for SARS-CoV-2 infection on Day -1.
10. Systolic BP in the range of 80 to 140 mmHg and diastolic BP in the range of 50 to 95 mmHg at Screening. If out of range, BP may be repeated once at the discretion of the Investigator.
11. Male or female

    * Male participants with partners of childbearing potential must agree to use contraception from Screening through at least 24 weeks after the last dose of study intervention and refrain from donating sperm during this period (see Section 10.4).
    * Female participants may not be pregnant or breastfeeding, and at least one of the following conditions must apply:

      * Is not a woman of childbearing potential (WOCBP) or
      * If a WOCBP, must agree to follow the contraceptive guidance (see Section 10.4), beginning at consent and the first Screening visit and for at least 24 weeks after the last dose of study intervention.
12. BMI within the range 18.0 to 32.0 kg/m2 (inclusive).
13. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

Exclusion Criteria:

History of any medical condition that may interfere with the metabolism of study intervention or with the clinical and laboratory assessments in this study. 2. History of serious, persistent medical conditions, including liver, gastrointestinal, pulmonary, renal, or cardiovascular abnormalities. 3. History of suicidal attempt at any time or an answer of "yes" on any of the following items in the C-SSRS at Screening:

1. Items 1 or 2 of the Suicidal Ideation section, if ideation occurred in the previous 12 months.
2. Items 4 or 5 of the Suicidal Ideation section, in lifetime.
3. Any item of the Suicidal Behavior section of the C-SSRS, in lifetime. 4. Any history of severe or recent clinically significant depression, anxiety, bipolar disorder, schizophrenia, or other neuropsychiatric disorder that, in the judgement of the Investigator, represents a safety risk to the participant were they to participate in the trial, as informed by the participant's medical history and/or responses to the MINI Screen Questionnaire. 5. History of substance use disorder (SUD) or illicit drug use (excluding cannabis) within the preceding 12 months. 6. History of alcohol withdrawal symptoms including delirium tremens or alcohol-related seizures. 7. Any condition that, in the opinion of the Investigator, would make the participant unsuitable for participation or could interfere with participation in or completion of the study, including:

a. Poorly controlled or unstable hypertension. b. Diabetes mellitus treated with insulin or hypoglycemic agents (including metformin) or HbA1C > 7%. Asthma requiring hospital admission within the preceding 12 months. NOTE: Persons with clinically stable asthma who have not been hospitalized in the prior year and are treated only with orally inhaled medications are not excluded. d. Currently poorly controlled endocrine conditions, except for hypothyroidism that is stable (no treatment change in prior 6 months). e. Significant infection or known systemic inflammatory process ongoing at Screening.

f. History of chronic or recurrent UTI, or UTI within 1 month prior to Screening.

8. History of malignancy within the preceding 5 years requiring treatment, with the exception of excised low grade basal cell skin neoplasms. 9. History of any concomitant medical condition for which alcohol consumption is prohibited or advised against by the participant's physician or health care provider.

10. SARS-CoV-2 infection in the 14 days prior to randomization. 11. Clinically significant illness within the 7 days prior to the first administration of study intervention. History of multiple drug allergies or a history of allergic reaction to an oligonucleotide based therapy.

13. Use of prescription medications (except for hormonal replacement/contraceptive medication for women and inhaled medication for treatment of clinically stable asthma) within 14 days or 5 half-lives (whichever is longer) prior to administration of study intervention. Participants being treated for hypothyroid disease must be on stable treatment (no treatment changes in the preceding 6 months). 14. Receipt of any vaccine (including COVID-19) within 14 days prior to the first administration of study intervention. 15. Regular use of OTC medications, including NSAID (periodic or occasional NSAID use to control temporary pain is not exclusionary). 16. Previously participated in Dicerna Study DCR-AUD-101. 17. Has received an investigational agent within 30 days or 5 half-lives (whichever is longer) prior to dosing or is in follow-up of another clinical study prior to initial dosing with the study intervention. 18. Clinically significant abnormalities in vital signs at Screening: pulse rate (< 40 bpm or > 90 bpm), respiratory rate, or temperature. 19. Clinically significant abnormalities in 12-lead ECG at Screening or predose on Day 1, including QTcF > 470 msec in females and > 450 msec in males. 20. Positive urine drug test at Screening or Day -1. Tests positive for cannabis are not exclusionary. 21. Seropositive for antibodies to HIV, HBV, or HCV at Screening (historical testing may be used if performed within the 3 months prior to screening). NOTE: In participants with previous treatment for hepatitis C with direct-acting HCV medication and seropositivity for HCV, or in participants with prior infection and spontaneous resolution, HCV RNA must be undetectable (at least 2 negative HCV RNA tests at least 12 weeks apart), and the HCV infection must have been resolved or cured > 3 years prior to initial dosing with the investigational medication. 22. Safety laboratory test result at Screening considered clinically unacceptable for study participation by the Investigator. 23. History of intolerance to SC injection(s) or significant abdominal scarring that could potentially hinder study intervention administration or evaluation of local injection site tolerability. 24. Scheduled for an elective surgical procedure during the conduct of this study.

25. Donation of > 500 mL of blood within the 2 months prior to administration of study intervention or donation of plasma within 7 days prior to Screening.

Life Style Considerations:

1. Study participants are to refrain from drinking alcohol for 24 hours prior to each EIA and must have a negative breath-alcohol test on the day of the study visit.
2. Study participants will be advised to avoid consuming more than 4 drinks during any drinking session outside of in-clinic EIAs.
3. Study participants will be instructed to stop drinking at the onset of any ethanol reaction symptoms during outside drinking sessions.
4. Tobacco/nicotine use is not restricted.
5. Study participants are to refrain from using cannabis for 24 hours prior to each EIA and must have a negative urine-drug test on the day of the study visit.
6. Study participants should abstain from strenuous exercise for 24 hours before each blood collection for clinical laboratory tests. Participants may participate in light recreational activities (e.g., walking at a pace < 3 miles per hour, shopping, watering plants) in that 24-hour time period.
7. For each EIA study visit, participants will be required to fast for at least 3 hours and then will be fed a standardized meal in the clinic prior to administration of ETOH for the EIA.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-01-29 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2023-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Hanrahan, MD, MPH, Study Director — Dicerna Pharmaceuticals, Inc., a Novo Nordisk company; Lev G. Gertsik, MD, Principal Investigator — Parexel
Locations (1):
- Parexel Los Angeles Early Phase Clinical Unit, Glendale, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 1 site in the United States of America.
Pre-assignment Details: In this trial total 16 healthy participants were randomized in 3:1 ratio to DCR-AUD or placebo.
Groups:
- DCR-AUD: Participant received DCR-AUD 480 mg, subcutaneous injection on Day 1, Day 29 and Day 57.
- Placebo: Participant received DCR-AUD matching placebo, subcutaneous injection on Day 1, Day 29 and Day 57.
Period: Overall Study
Arm/Group | DCR-AUD | Placebo
Started | 12 | 4
Pharmacokinetic Population | 12 | 0
Pharmacodynamic Population | 12 | 4
Completed | 12 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population (SP): All participants randomized to study intervention and who receive at least 1 dose of DCR-AUD or placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | DCR-AUD | Placebo | Total
Number analyzed (Participants) | 12 | 4 | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.3 (9.91) | 38.0 (3.37) | 39.0 (8.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 1 | 10
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 6
  Not Hispanic or Latino | 7 | 3 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 9 | 2 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An Adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention. A TEAE is defined as an AE that begins or that worsens in severity after the study drug has been administered. An SAE is defined as any untoward medical occurrence that at any dose: results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, leads to a congenital anomaly /birth defect, is the other important medical event.
Time Frame: From Day 1 up to 24 Weeks
Population: SP: All participants randomized to study intervention and who receive at least 1 dose of DCR-AUD or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | DCR-AUD | Placebo
Number analyzed (Participants) | 12 | 4
Participants
  TEAEs | 11 | 3
  SAEs | 0 | 0

2. Primary Outcome: Number of Participants With Severity Grades of TEAEs
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. A TEAE is defined as an AE that begins or that worsens in severity after the study drug has been administered. As per the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0, Grade 1: mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; treatment not indicated; Grade 2: moderate; minimal, local, or noninvasive treatment indicated; limiting age-appropriate activities of daily living; Grade 3: severe or medically significant but not immediately lifethreatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living; Grade 4: life-threatening consequences; urgent treatment indicated; Grade 5: fatal.
Time Frame: From Day 1 up to 24 Weeks
Population: SP: All participants randomized to study intervention and who receive at least 1 dose of DCR-AUD or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | DCR-AUD | Placebo
Number analyzed (Participants) | 12 | 4
Participants
  Grade 1 | 11 | 3
  Grade 2 | 3 | 0
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0

3. Primary Outcome: Number of Participants With Change From Baseline in Clinically Significant Abnormal Vital Signs
Description: Number of participants with change from baseline in clinically significant abnormal vital signs (temperature, pulse rate, respiratory rate, and blood pressure) is presented.
Time Frame: From Baseline (Day -1) up to 24 weeks
Population: SP: All participants randomized to study intervention and who receive at least 1 dose of DCR-AUD or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | DCR-AUD | Placebo
Number analyzed (Participants) | 12 | 4
Participants | 0 | 0

4. Primary Outcome: Number of Participants With Change From Baseline in Clinically Significant Abnormal Electrocardiogram (ECG)
Description: Number of participants with change from baseline in clinically significant abnormal ECG findings (Heart rate, PR interval, QRS interval, QT interval and QT interval using Fridericia's correction [QTcF]) is presented.
Time Frame: From Baseline (Day -1) up to 24 weeks
Population: SP: All participants randomized to study intervention and who receive at least 1 dose of DCR-AUD or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | DCR-AUD | Placebo
Number analyzed (Participants) | 12 | 4
Participants | 0 | 0

5. Primary Outcome: Number of Participants With Change From Baseline in Clinically Significant Abnormal Laboratory Values
Description: Number of participants with change from baseline in clinically significant abnormal laboratory values (hematology, clinical chemistry, coagulation and routine urinalysis parameters) is presented.
Time Frame: From Baseline (Day -1) up to 24 weeks
Population: SP: All participants randomized to study intervention and who receive at least 1 dose of DCR-AUD or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | DCR-AUD | Placebo
Number analyzed (Participants) | 12 | 4
Participants | 0 | 0

6. Primary Outcome: Number of Participants With Change From Baseline in Clinically Significant Physical Examination Findings
Description: Number of participants with change from baseline in clinically significant physical examination findings (assessments of the cardiovascular, respiratory, gastrointestinal, neurological, and skin systems and inspection of the injection site) is presented.
Time Frame: From Baseline (Day -1) up to 24 weeks
Population: SP: All participants randomized to study intervention and who receive at least 1 dose of DCR-AUD or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | DCR-AUD | Placebo
Number analyzed (Participants) | 12 | 4
Participants | 0 | 0

7. Secondary Outcome: Six Symptom Responses During Ethanol Interactions Assessments (EIAs)
Description: The degree of aldehyde dehydrogenase 2 (ALDH2) reduction was measured by quantitative assessment of 6 symptom (flushing, headache, palpitations, light-headedness, nausea, and vomiting) responses during EIAs. Each of 6 symptoms was assessed at each of the 4 time points during each EIA. Composite score at each time point was the sum of severity ratings for each of the 6 symptoms. Peak composite score (of the 3 post-alcohol initiation composite scores at each EIA test) was used as the subject's peak score for that EIA test. The point system was as follows: 0 point = symptom not present, 1 point = mild severity of symptom, 2 points = moderate severity of symptom and 3 points = severe severity of symptom. Participants were given a composite score, which was the sum of the scores of all 6 symptoms (highest possible score is 18).
Time Frame: Day -1 (baseline), Day 14, Day 28, Day 42, Day 56, Day 70, Day 84, Day 112, Day 140 and Day 168
Population: Pharmacodynamic Population (PP): All participants randomized to study intervention and who receive at least 1 dose of DCR-AUD or placebo and have at least 1 postdose PD assessment. Here, number analysed signifies participants with available data for each specified timepoints.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | DCR-AUD | Placebo
Number analyzed (Participants) | 12 | 4
Score on a scale
  Day -1 (baseline) | 0.3 (0.65) | 0.5 (0.58)
  Day 14 | 0.4 (0.67) | 0 (0)
  Day 28 | 0.8 (0.75) | 0.5 (0.58)
  Day 42 | 0.9 (1.08) | 0.8 (0.96)
  Day 56: number analyzed (Participants) | 11 | 4
  Day 56 | 1.1 (1.14) | 0.3 (0.50)
  Day 70 | 1.0 (1.21) | 0 (0)
  Day 84 | 1.1 (1.24) | 0 (0)
  Day 112: number analyzed (Participants) | 11 | 4
  Day 112 | 0.9 (1.22) | 0 (0)
  Day 140 | 0.8 (1.06) | 0.3 (0.50)
  Day 168 | 0.8 (0.87) | 0.3 (0.50)

8. Secondary Outcome: AUC0-last: Area Under the Plasma Concentration Curve From Time Zero to the Last Quantifiable Concentration of DCR-AUD
Description: AUC0-last is defined as the area under the plasma concentration curve from time zero to the last quantifiable concentration of DCR-AUD.
Time Frame: Day 1, Day 29 and Day 57
Population: Pharmacokinetic Population (PKP): All participants randomized to study intervention and who receive at least 1 dose of DCR-AUD and have at least 1 postdose PK assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per millilitre (h*ng/ mL)
Arm/Group | DCR-AUD
Number analyzed (Participants) | 12
hour*nanogram per millilitre (h*ng/ mL)
  Day 1 | 44100 (16.3)
  Day 29 | 41000 (16.9)
  Day 57 | 66200 (27.0)

9. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration of DCR-AUD
Description: Cmax is defined as maximum observed plasma concentration of DCR-AUD is presented.
Time Frame: Day 1, Day 29 and Day 57
Population: PKP: All participants randomized to study intervention and who receive at least 1 dose of DCR-AUD and have at least 1 postdose PK assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per millilitre (ng/mL)
Arm/Group | DCR-AUD
Number analyzed (Participants) | 12
nanogram per millilitre (ng/mL)
  Day 1 | 2530 (28.1)
  Day 29 | 2280 (32.3)
  Day 57 | 1900 (26.3)

10. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration of DCR-AUD (Cmax)
Description: Tmax is defined as time to reach the maximum plasma concentration (Cmax) of DCR-AUD.
Time Frame: Day 1, Day 29 and Day 57
Population: as for outcome 9
Measure: Median (Full Range); unit: Hours
Arm/Group | DCR-AUD
Number analyzed (Participants) | 12
Hours
  Day 1 | 4.95 [1.00 to 8.01]
  Day 29 | 4.99 [1.02 to 8.00]
  Day 57 | 3.98 [1.00 to 8.10]

11. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration of Acetaldehyde
Description: Maximum observed plasma concentration of acetaldehyde levels was measured to evaluate the pharmacodynamic effects of ALDH2 reduction by DCR-AUD during serial EIAs.
Time Frame: Day -1 (baseline), Day 14, Day 28, Day 42, Day 56, Day 70, Day 84, Day 112, Day 140 and Day 168
Population: PP: All participants randomized to study intervention and who receive at least 1 dose of DCR-AUD or placebo and have at least 1 postdose PD assessment. Here, number analysed signifies participants with available data for each specified timepoints.
Measure: Mean (Standard Deviation); unit: Micromolar (μM)
Arm/Group | DCR-AUD | Placebo
Number analyzed (Participants) | 12 | 4
Micromolar (μM)
  Day -1 (baseline): number analyzed (Participants) | 11 | 3
  Day -1 (baseline) | 19.8 (5.71) | 28.3 (17.1)
  Day 14: number analyzed (Participants) | 12 | 3
  Day 14 | 21.6 (14.1) | 24.3 (3.51)
  Day 28 | 40.2 (27.9) | 15.1 (6.88)
  Day 42: number analyzed (Participants) | 12 | 3
  Day 42 | 34.0 (19.9) | 12.6 (3.51)
  Day 56: number analyzed (Participants) | 11 | 3
  Day 56 | 53.9 (29.6) | 26.7 (14.9)
  Day 70: number analyzed (Participants) | 12 | 3
  Day 70 | 58.6 (46.3) | 36.3 (23.8)
  Day 84 | 62.9 (23.0) | 20.7 (13.8)
  Day 112: number analyzed (Participants) | 11 | 4
  Day 112 | 80.3 (37.8) | 25.3 (21.7)
  Day 140 | 98.3 (40.7) | 21.9 (16.2)
  Day 168 | 132 (48.6) | 30.6 (24.1)

12. Secondary Outcome: AUC0-4: Area Under the Concentration Time Curve From Time 0 to Fixed Time 4 of Acetaldehyde
Description: Area under the concentration time curve from time 0 to fixed time 4 of acetaldehyde levels was measured to evaluate the pharmacodynamic effects of ALDH2 reduction by DCR-AUD during serial EIAs.
Time Frame: Day -1, Day 14, Day 28, Day 42, Day 56, Day 70, Day 84, Day 112, Day 140 and Day 168
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Micromolar*hours (μM*h)
Arm/Group | DCR-AUD | Placebo
Number analyzed (Participants) | 12 | 4
Micromolar*hours (μM*h)
  Day -1: number analyzed (Participants) | 11 | 3
  Day -1 | 47.8 (20.3) | 65.8 (48.0)
  Day 14: number analyzed (Participants) | 12 | 3
  Day 14 | 48.2 (43.1) | 62.1 (11.6)
  Day 28 | 93.2 (68.6) | 32.0 (24.6)
  Day 42: number analyzed (Participants) | 12 | 3
  Day 42 | 81.8 (52.9) | 21.6 (10.7)
  Day 56: number analyzed (Participants) | 11 | 3
  Day 56 | 131 (81.8) | 54.4 (48.9)
  Day 70: number analyzed (Participants) | 12 | 3
  Day 70 | 135 (88.9) | 78.3 (51.2)
  Day 84 | 135 (52.4) | 49.5 (45.6)
  Day 112: number analyzed (Participants) | 11 | 4
  Day 112 | 187 (75.9) | 57.5 (63.6)
  Day 140 | 228 (85.1) | 56.8 (63.5)
  Day 168 | 334 (93.9) | 69.4 (70.0)

13. Secondary Outcome: Change From Baseline in Heart Rate
Description: Heart rate is measured to evaluate the PD effects of ALDH2 reduction by DCR-AUD during serial EIA. Heart rate was monitored by telemetry during the EIAs.
Time Frame: Baseline, Day 169
Population: SP: All participants randomized to study intervention and who receive at least 1 dose of DCR-AUD or placebo.
Measure: Mean (Standard Deviation); unit: beats per minute (beats/min)
Arm/Group | DCR-AUD | Placebo
Number analyzed (Participants) | 12 | 4
beats per minute (beats/min) | 1.9 (9.09) | 4.3 (8.10)

14. Secondary Outcome: Change From Baseline in Facial Skin Temperature
Description: Change in facial skin temperature was measured to evaluate the PD effects of ALDH2 reduction by DCR-AUD during serial EIAs.
Time Frame: Baseline, Day 169
Population: SP: All participants randomized to study intervention and who receive at least 1 dose of DCR-AUD or placebo.
Measure: Mean (Standard Deviation); unit: degree celsius
Arm/Group | DCR-AUD | Placebo
Number analyzed (Participants) | 12 | 4
degree celsius | -0.05 (0.555) | 0.03 (0.704)

ADVERSE EVENTS:
Time Frame: From Day 1 until end of the study (24 weeks)
Description: Safety Population (SP): All participants randomized to study intervention and who receive at least 1 dose of DCR-AUD or placebo. All serious and non-serious adverse events presented here are treatment emergent adverse events.
Arm/Group | DCR-AUD | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/4
Other Adverse Events (participants affected / at risk) | 11/12 | 3/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DCR-AUD (N=12) | Placebo (N=4)
Headache (Nervous system disorders) | 6 (27) | 0 (0)
Dizziness (Nervous system disorders) | 3 (7) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 5 (8) | 0 (0)
Hot flush (Vascular disorders) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (8) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0)
Palpitations (Cardiac disorders) | 3 (4) | 0 (0)
Injection site bruising (General disorders) | 2 (2) | 0 (0)
Injection site erythema (General disorders) | 2 (2) | 0 (0)
Injection site discolouration (General disorders) | 1 (1) | 0 (0)
Injection site dryness (General disorders) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property

DOCUMENTS (2):
  • Study Protocol (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/98/NCT05845398/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT05845398/SAP_001.pdf